CLINICAL TRIAL: NCT05922956
Title: Facial Emotion Recognition in Patients With Euthymic Bipolar Disorder I and II
Acronym: REF-BIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier le Vinatier (Unknown); Pôle Ressource Évaluation et Réhabilitation Psycho-sociale, EPSM de l'Oise (Unknown); Centre de santé mentale MGEN (Unknown); Centre Hospitalier Philippe Pinel, Amiens (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0009
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Social Cognition; Facial Emotion Recognition; Facial Affect; Bipolar Disorder I and II
Keywords: social cognition; facial emotion recognition; facial affect; bipolar disorder I and II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with bipolar disorder 1 (Experimental)
  Interventions: Other: Facial emotion recognition test
- patients with bipolar disorder 2 (Experimental)
  Interventions: Other: Facial emotion recognition test
- healthy controls (Active Comparator)
  Interventions: Other: Facial emotion recognition test

INTERVENTIONS:
Other: Facial emotion recognition test — Facial emotion recognition test (TREF), questionnaires including self-administered questionnaires

SUMMARY:
The facial emotion recognition is a basic social skill for successful social interactions. Several meta-analyses and recent studies found impairments of the perception of facial emotions in patients with euthymic bipolar disorder. Few studies compared recognition of facial emotions impairments during euthymia in patients with bipolar disorder type 1 and 2. These studies included low population samples (N<60). There were discrepancies in results of these studies. Szanto suggested that facial emotion recognition impairments were correlated with suicidal risk and social isolation. These impairments should be taking into account regarding psycho-social treatments in patients with bipolar disorder.

This study aims to evaluate facial emotion recognition in patients with bipolar I and II disorders compared to healthy controls, using the facial emotion recognition test (TREF). The objective of the present study is to compare TREF scores in a group of patients with bipolar 1, a group of patients with bipolar 2 disorder and a group with healthy controls. In addition, the investigators will investigate the relationships between TREF scores and levels of self-esteem and mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Patient group :
* Male or female patients, between 18 and 60 years old
* Diagnosis of Bipolar Disorder I or Bipolar Disorder II according to DSM-IV criteria, using the French version of the Mini-International Neuropsychiatric Interview (MINI)
* Strictly euthymic defined by Hamilton Depression Rating Scale (17 items) ≤ 5 and Young Mania Rating Scale ≤ 5 for at least two months.
* Native French speakers
* Affiliated to the French social security system
* Giving their written informed consent

Control group :

* Male or female control subjects, aged between 18 and 60 years old, assessed using TREF
* Native French speakers
* Giving their written informed consent

Exclusion Criteria:

* Patient group :
* History of mental retardation assessed by the French version of the National Adult Reading Test
* Neurological illness or any clinical condition that could affect cognitive performance (history of head injury with loss of consciousness lasting more than 5 minutes multiple sclerosis, stroke etc.)
* Electroconvulsive therapy within the last 6 months
* Alcohol and Drug dependence (except tobacco and caffeine) according to DSM-IV criteria using the French version of the Mini-International Neuropsychiatric Interview (MINI).
* Learning disability or difficulty with fluent use of the French language
* Patient with mandatory care
* Long-Term use of non-psychotropic medication with psychotropic effects (opiates, Baclofen)

Control group :

* History of mental retardation estimated by the French version of the National Adult Reading Test
* Neurological illness or any clinical condition that could affect cognitive performance (history of head injury with loss of consciousness lasting more than 5 minutes multiple sclerosis, stroke etc.)
* Current Mood disorder/ Lifetime Psychotic Disorder according to DSM-IV criteria using the French version of the Mini-International Neuropsychiatric Interview (MINI)
* Neither history of psychotic or affective disorders in a first-degree family member
* Alcohol and Drug dependence (except tobacco and caffeine) according to DSM-IV criteria using the French version of the Mini-International Neuropsychiatric Interview (MINI)
* Learning disability or difficulty with fluent use of the French language
* Long-Term use of non-psychotropic drugs with psychotropic effects (opiates, Baclofen) and psychotropic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
variation of TREF scores in tree groups of subjects | 16 months
  TREF scores in tree groups of subjects (group of patients with bipolar disorder 1, group of patients with bipolar disorder 2 and group of healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No